CLINICAL TRIAL: NCT06697600
Title: A Decisional Intervention for Older Adults With Acute Myeloid Leukemia and Their Caregivers
Acronym: UR-GOAL RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor, Division of Hematology/Oncology, Department of Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UOCPC24064; 1R01CA288318-01A1 (NIH)
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Oncology; Myeloid Leukemia, Acute; Cancer
Keywords: older adults; geriatric oncology; caregivers
MeSH Terms: conditions — Neoplasms; Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to either the UR-GOAL arm or the attention control arm. If the patient has a caregiver that agrees and consents to participate in the study, the caregiver will be enrolled onto the same arm as the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UR-GOAL Intervention (Experimental): Patients will view an AML video, complete the best-worst scaling, and be provided with a summary report consisting of their priorities; they will will be asked to review and discuss at upcoming clinical visits. Caregivers, if available, will view the same AML video and be provided with the same summary report. Oncologists will be provided with a summary report consisting of the patient's geriatric assessment, priorities, and perception of prognosis; they will be asked to review and discuss at upcoming clinical visits.
  Interventions: Behavioral: UR-GOAL
- Attention Control Arm (No Intervention): Patients will view a nutritional video, complete a nutrition questionnaire, and will be provided with a nutrition handout and asked to review and discuss at upcoming clinical visits. Caregivers, if available, will view the nutritional video, and will be provided with a nutrition handout and asked to review and discuss at upcoming clinical visits. Oncologists will be provided with the patient's completed nutrition questionnaire and asked to review and discuss at upcoming clinical visits.

INTERVENTIONS:
Behavioral: UR-GOAL — Patients will view an AML video, complete the best/worst scaling, will be provided with a summary report, and will be asked to review and discuss at upcoming clinical visits. Caregivers, if available, will view an AML video, will be provided with a summary report, and will be asked to review. Oncologists will be provided with a summary report and will be asked to review and discuss at upcoming clinical visits.
  Arms: UR-GOAL Intervention

SUMMARY:
This is a multicenter randomized controlled trial that assesses the efficacy of a decisional intervention [University of Rochester-Geriatric Oncology assessment for Acute myeloid Leukemia (UR-GOAL)] compared to an attention control.

DETAILED DESCRIPTION:
This is a multicenter randomized controlled trial with four sites that assesses the efficacy of a decisional intervention [University of Rochester-Geriatric Oncology assessment for Acute myeloid Leukemia (UR-GOAL)] compared to an attention control. Subjects will be randomized 1:1 to either the intervention arm or the attention control arm. Compared to an attention control, UR-GOAL will improve patient distress, observed and patient-perceived shared decision making (SDM), and patient decisional conflict.

ELIGIBILITY:
Patients

Inclusion criteria:

* Age ≥60 years (from date of consent, confirmed on electronic medical records)
* A new diagnosis of AML

  * Diagnosis can be based on the International Consensus Classification or World Health Organization
  * Myeloid sarcoma is allowed
  * AML with central nervous system involvement is allowed
* Cancer-directed treatment has not started

  * Treatment to temporarily decrease white blood cells is acceptable; these may include hydroxyurea, leukapheresis, or cytarabine
  * Intrathecal chemotherapy is acceptable
* The patient's oncologist has been or will be enrolled on the study
* English or Spanish-speaking
* Patients without a caregiver will still be eligible to participate in the study Exclusion criteria
* A diagnosis of acute promyelocytic leukemia
* Patients with psychiatric or cognitive conditions which the treating oncologist believes prohibits informed consent or compliance with study procedures
* Prior cancer-directed treatment for AML

Caregivers

Inclusion criteria:

* Selected by the patient when asked if there is a "family member, partner, friend or caregiver [age 18 or older] with whom you discuss or who can be helpful in healthrelated matters."
* Caregiver may be paid/professional or informal caregiver
* Able to provide informed consent
* English or Spanish-speaking

Oncologists

Inclusion criteria:

• Oncologists caring for patients with AML Exclusion criteria

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Distress Thermometer Questionnaire at 1 month | 1 month
  A self-report measure to capture distress and identify a list of sources of that distress. This is a 10-item scale, rated from 0-10 (0=no distress, 10=severe distress), with a possible total of 10; a higher score indicates greater distress.

SECONDARY OUTCOMES:
9-item Shared Decision Making Questionnaire at 2 weeks | 2 weeks
  9-item Shared Decision Making Questionnaire at 2 weeks
Decisional Conflict Scale Questionnaire at 2 weeks | 2 weeks
  Decisional Conflict Scale Questionnaire at 2 weeks
Observed shared decision making | Day 0
  OPTION5 instrument from audio-recorded treatment decision-making clinical visits

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Division of Hematology and Oncology, Birmingham, Alabama
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Section of Hematology/Oncology, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LoCastro M, Sanapala C, Wang Y, Jensen-Battaglia M, Wittink M, Norton S, Klepin HD, Richardson DR, Mendler JH, Liesveld J, Huselton E, O'Dwyer K, Cortes AM, Rodriguez C, Dale W, Loh KP. Patient-centered communication tool for older patients with acute myeloid leukemia, their caregivers, and oncologists: A single-arm pilot study. Cancer Med. 2023 Apr;12(7):8581-8593. doi: 10.1002/cam4.5547. Epub 2022 Dec 19. PMID 36533397